CLINICAL TRIAL: NCT01724788
Title: Pharmacokinetic Profile and Pharmacodynamic Characteristics of a Furosemide High Dosage Formulation (PRLasix® Special, Tablets 500 mg) in Patients With Chronic Renal Failure Undergoing Peritoneal Dialysis
Brief Title: Pharmacokinetic Profile and Pharmacodynamic Characteristics of a Furosemide High Dosage Formulation in Patients With Chronic Renal Failure Undergoing Peritoneal Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FUROSL06121; U1111-1127-0839 (Other: UTN)
Record Dates: First submitted 2012-10-30; First posted 2012-11-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide PO - IV (Experimental): Oral furosemide allocated at the beginning of Period 1, then cross-over to IV furosemide (a minimum 7-day diuretic free washout period required between the two periods)
  Interventions: Drug: FUROSEMIDE; Drug: FUROSEMIDE (HOE058)
- Furosemide IV - PO (Experimental): IV furosemide allocated at the beginning of Period 1, then cross-over to oral furosemide (a minimum 7-day diuretic free washout period required between the two periods)
  Interventions: Drug: FUROSEMIDE; Drug: FUROSEMIDE (HOE058)

INTERVENTIONS:
Drug: FUROSEMIDE — Pharmaceutical form: Solution Route of administration: Intravenous
  Other Names: Furosemide Special Injection
Drug: FUROSEMIDE (HOE058) — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: Lasix® Special

SUMMARY:
Primary Objective:

* To determine the absolute bioavailability of furosemide 500 mg (Lasix® Special) oral formulation in patients with chronic renal failure undergoing peritoneal dialysis.

Secondary Objectives:

* To determine the pharmacokinetic profiles of furosemide 500 mg (Lasix® Special) oral formulation and 250 mg IV formulation
* To compare the pharmacodynamic characteristics of furosemide 500 mg (Lasix® Special) oral formulation and 250 mg IV formulation

DETAILED DESCRIPTION:
* Screening: 7 to 10 days
* Treatment period: 14 days (Period 1: 7 days; Period 2: 7 days)
* End of study: 7 days after the last dosing,
* Total duration from screening per subject: 22 to 25 days.

ELIGIBILITY:
Inclusion criteria :

* Male or female, 18 years old or older, with chronic renal failure undergoing peritoneal dialysis for at least 3 months.
* Women of childbearing age should have a negative pregnancy test before administration of the study drug

Exclusion criteria:

* Contra-indications to furosemide, including:

  * Hypersensitivity to furosemide or to sulphonamide-derived drugs or to any ingredient in the formulation or component of the container.
  * Glomerular filtration rate below 5 mL/min
  * Glomerular filtration rate above 20 mL/min
  * Severe liver disease
  * Patients with renal failure accompanied by hepatic coma and precoma
  * Renal failure due to poisoning with nephrotoxic or hepatotoxic substances
  * Severe hyponatremia, hypokalemia, hypovolemia, dehydration or hypotension
  * Nursing women
* Pregnancy
* Treatment with any diuretic, which cannot be discontinued with the required washout period before the first drug administration
* Existence of any surgical or medical condition, which, in the judgment of the clinical investigator, might interfere with absorption, distribution, metabolism or excretion of drugs.
* Psychiatric or cognitive disturbance or illness, or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect patient safety and/or compliance.
* Treatment with the following inhibitors of secretion at the renal level: clarithromycin, erythromycin, itraconazole, cyclosporin, ketoconazole, quinidine, and verapamil, which cannot be discontinued during the course of the study.

Interfering substance:Subjects must abstain from alcohol and beverages containing stimulating xanthine derivates (e.g. coffee and tea) during the entire study period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) of a single 500-mg oral tablet | Day 1, 4, 8, 11

SECONDARY OUTCOMES:
To determine the pharmacokinetic parameters of furosemide (po and iv) measured by Cmax (maximum (peak) plasma drug concentration) after single dose administration | Day 1, 4, 8, 11
To determine the pharmacokinetic parameters of furosemide (po and iv) measured by Tmax (time to reach peak or maximum concentration) following drug administration | Day 1, 4, 8, 11
To determine the pharmacokinetic parameters of furosemide (po and iv) measured by AUCT 0-72 (area under curve from the time zero to 72h) | Day 1, 4, 8, 11
To determine pharmacodynamic characteristics of furosemide (po and iv) including the excretion against time of urinary volume, urinary excretion, urea and creatinine | 0, 6, 12, 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 124002, Montreal, Canada